CLINICAL TRIAL: NCT01039805
Title: A Double-blind, Randomized, Placebo Controlled Phase II Study to Evaluate the Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of Single Doses of the Oral Motilin Receptor Agonist GSK962040, in Critically Ill Male and Female Patients With Enteral Feed Intolerance
Brief Title: Evaluation of Single Doses of GSK962040 in Critically Ill Patients With Enteral Feed Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112571
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Gastroparesis
Keywords: GSK962040; 13C octanoic acid breath test; pharmacokinetics; critically ill patients; gut motility; pharmacodynamics; tolerability; single dose; gastric emtpying
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects randomized to either GSK962040 (50 mg) or placebo
  Interventions: Drug: GSK962040 (50 mg); Drug: Placebo
- Cohort 2 (Experimental): Subjects randomized to either GSK962040 (75 mg) or placebo
  Interventions: Drug: Placebo; Drug: GSK962040 (75 mg)

INTERVENTIONS:
Drug: GSK962040 (50 mg) — Cohort 1 = 50 mg
  Arms: Cohort 1
Drug: Placebo — matching placebo
Drug: GSK962040 (75 mg) — Cohort 2 = 75 mg
  Arms: Cohort 2

SUMMARY:
The aims of MOT112571 are to assess the pharmacodynamic effects, safety, tolerability, pharmacokinetics, and potential therapeutic benefit of single doses of GSK962040 in critically ill patients with delayed gastric emptying and who are intolerant to enteral feeding.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-85 years of age, at the time consent is obtained.
* Mechanically ventilated on the Intensive Care Unit who has become intolerant of nasogastric enteral feeding.
* intolerance of nasogastric tube feeding is defined as a gastric aspirate volume (GRV) >250 mL at least 6 hours after commencing feeding at >40 mL/hr.
* Expected to remain mechanically ventilated for at least 48 hours after enrollment and expected to survive for at least 24 hours post dose of study medication.
* Subject has a nasogastric tube for enteral feeding.
* Body weight > or = 50 kg
* Written informed consent may be obtained from a legally acceptable representative, which includes compliance with the requirements and restrictions listed in the consent form. In most cases, consent will be sought from next of kin as the subject will not be competent to give their own consent.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST and ALT < 3xULN; alkaline phosphatase and bilirubin < or = 2xULN.
* Subjects who have rapidly rising aminotransferases or for whem there is not a plausible explanation for the observed elevation will not be enrolled
* LFTs will be checked for eligibility on screening and again prior to dosing with GSK962040.

Exclusion Criteria:

* Subjects that have received a gastric prokinetic agent in the previous 24 h (e.g., erythromycin, azithromycin, metoclopramide). These agents are prohibited for the duration of the study.
* Subjects whose clinical condition is deteriorating rapidly or any subject for whom the investigator does not consider there is a reasonable expectation that they will be able to complete the study.
* Subjects who are known to be infected with Hepatitis B, Hepatitis C, or HIV viruses.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prohibited medications listed in Section 9.2 within the restricted timeframe relative to dosing of study medication.
* Subjects with renal failure requiring replacement therapy (dialysis or filtration).
* Subjects for whom the reason for admission to ICU was an overdose (deliberate or accidental; medicinal product or not).
* Subjects with altered upper gastrointestinal tract anatomy and subjects who have undergone upper gastrointestinal tract surgery on this admission to ICU.
* Subjects with bowel obstruction or perforation.
* Subject has a gastric pacemaker
* Subject is receiving parenteral feeding
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 3 days
Safety and tolerability of GSK962040 | 5 days
Pharmacokinetic parameters of GSK962040: Cmax, Tmax, AUC(0-inf), AUC(0-t), CL/F, V/F, and half-life | 3 days

SECONDARY OUTCOMES:
Pre and post GSK962040 dose Gastric Residual Volume (GRV) | Duration of dosing
Pharmacokinetic parameters of paracetamol | duration of dosing
Pharmacokinetic parameters of 3OMG | duration of dosing
Plasma concentrations of motilin | duration of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chapman MJ, Deane AM, O'Connor SL, Nguyen NQ, Fraser RJ, Richards DB, Hacquoil KE, Vasist Johnson LS, Barton ME, Dukes GE. The effect of camicinal (GSK962040), a motilin agonist, on gastric emptying and glucose absorption in feed-intolerant critically ill patients: a randomized, blinded, placebo-controlled, clinical trial. Crit Care. 2016 Aug 1;20(1):232. doi: 10.1186/s13054-016-1420-4. PMID 27476581
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112571 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register